CLINICAL TRIAL: NCT03310697
Title: Toxicological Screening by GC-MS Among Children Admitted for a First Afebrile Seizure (CASTox): a Pilot Study
Brief Title: Toxicological Screening by GC-MS Among Children Admitted for a First Afebrile Seizure
Acronym: CASTox
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RC31/16/8246; 2017-A01319-44 (Other: IDRCB)
Record Dates: First submitted 2017-07-20; First posted 2017-10-16 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Afebrile Seizure (Finding)
Keywords: Afebrile seizure; Toxicological screening; Chromatography; Mass spectrometry; Children
MeSH Terms: conditions — Signs and Symptoms | interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: Transverse prevalence study. For each child, a toxicological screening will be carried out on the blood and urine for the research of proconvulsive molecules by conventional technique on the one hand and by gas chromatography coupled with a mass spectrograph on the other hand.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with afebrile seizure (Experimental): For each child, a toxicological screening will be carried out on the blood and urine for the research of proconvulsive molecules by conventional technique on the one hand and by gas chromatography coupled with a mass spectrograph on the other hand.
  Intervention : Collection of blood and urine samples, and Clinical examination
  Interventions: Other: Collection of blood and urine samples; Other: Clinical examination

INTERVENTIONS:
Other: Collection of blood and urine samples — For each child, a toxicological screening will be carried out on the blood and urine for the research of proconvulsive molecules by conventional technique on the one hand and by gas chromatography coupled with a mass spectrograph on the other hand.
Other: Clinical examination — The other clinical data, any other biological samples or additional examinations are done under the opinion of the clinician or the neuropediatrics.

SUMMARY:
Before the age of 14 years, 1% of the paediatric population will develop a seizure. The only systematically required complementary examination is an electroencephalogram (EEG). Additional biological or radiological examinations depend on the circumstances, the past medical history of the patient and other associated symptoms or clinical signs. A seizure can be the first sign of acute intoxication and represents a severity criterion. Failure to detect the toxic cause of a seizure can lead to a delay in the access or administration of an antidote if applicable. This can lead to target organ toxicity due to the absence of specific treatment. In the current French guidelines for a first seizure, a toxicological analysis is recommended if there is a possibility of exposure to toxic medications or products. However, this screening is often missing, unless a witness suggests that the child may have been exposed to a toxin.The recognition of a paediatric toxidrome is low among paediatricians, paediatric neurologists or emergency physicians. This is due to a lack of knowledge in clinical toxicology and the screening for toxic aetiology is not frequently or irrelevantly prescribed. There is an increasing number of proconvulsive molecules on the market. These molecules are not targeted in classic toxic screening. As result, a toxic cause of a seizure may be missed unless specific screening is performed. For all these reasons, little is known about the prevalence of toxic causes after a first episode of non-febrile seizure and probably under estimated in the paediatric population, especially in young children. New technologies for toxic detection like chromatography combined with mass spectrometry allow wide screening on different matrix. Initially dedicated to forensic analysis, they are more widely accessible for the exploration of the patients. The CASTox study is based on this context.

The first aim will be to evaluate the prevalence of a toxicological cause by a systematic blood and urine screening of children admitted to Toulouse paediatric emergency unit for a first afebrile seizure. Moreover, secondary aim will be to describe the effect of the systematic screening on the management of the children.

DETAILED DESCRIPTION:
Before the age of 14 years, 1% of the paediatric population will develop a seizure. The only systematically required complementary examination is an electroencephalogram (EEG). Additional biological or radiological examinations depend on the circumstances, the past medical history of the patient and other associated symptoms or clinical signs. A seizure can be the first sign of acute intoxication and represents a severity criterion. Failure to detect the toxic cause of a seizure can lead to a delay in the access or administration of an antidote if applicable. This can lead to target organ toxicity due to the absence of specific treatment. In the current French guidelines for a first seizure, a toxicological analysis is recommended if there is a possibility of exposure to toxic medications or products. However, this screening is often missing, unless a witness suggests that the child may have been exposed to a toxin.The recognition of a paediatric toxidrome is low among paediatricians, paediatric neurologists or emergency physicians. Since the end of the 90s, the molecules usually incriminated with seizure onset after intoxication are: with a high risk (polycyclic antidepressant, theophylline, isoniazid); intermediate risk (fluoroquinolones, tramadol, lidocaine, lithium, anticonvulsive medications) and low risk (selective serotonin reuptake inhibitors). Among infants, the molecules are quite different mainly because of the unintentional or malicious aspect of the intoxication and are dominated by sympathomimetic agents, antihistamine drugs, anticholinergic molecules, antidepressants and muscle relaxants. New drugs have been associated with seizures in young intoxicated children like bupropion, tramadol and venlafaxine. These agents are not detected by usual toxic analysis.

For each patient and after getting the signed consent form, a toxicological analysis will be performed on blood and urine samples to extensively screen for proconvulsive molecules (alcohols, polycyclic antidepressants, salicylates, anticonvulsive medications (carbamazepine, phenytoin, valproic acid), drugs (cocaine and its metabolites, amphetamines, methamphetamine (ecstasy), cannabis, buprenorphine, methadone, mephedrone, codeine, pholcodine, hydromorphone), benzodiazepines, caffeine, theophylline, lidocaine, isoniazid, mefenamic acid, tramadol, ephedrine).

This analysis will be performed using classic approach (immunoenzymatic detection) and by chromatography (GC) associated to mass spectrometry (MS) (Laboratory of Toxicology, University Hospital of Toulouse) - The other clinical data, biological results or tests requested by the physician in charge will be reported from the computerized medical file of each patient.

For each patient hospitalized, a follow-up visit will be scheduled during hospitalization in order to report management of the children.

ELIGIBILITY:
Inclusion Criteria:

* Being aged between 1 month and 15 years for boys and 1 month and 11 years for girls
* Any first episode of afebrile seizure, independent of duration, type (generalized or not) occurring in children without any previous neurological history and admitted to Toulouse level III paediatric emergency unit (University Children Hospital, Toulouse)
* Consent form signed by parents or legal guardian

Exclusion Criteria:

* Patient transferred from another hospital
* Absence of consent form signed by parents or legal guardian
* Seizure in a febrile context at the moment of inclusion
* Known history of neurological disorders
* Any kind of diagnosed epilepsy
* Renal or hepatocellular insufficiency
* Recent head trauma
* Coagulation disorders (hemophilia, secondary or primary thrombopenia)
* Known exposure to toxic molecules

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
Detection of one or several toxic molecules. | Day 1
  Analyzed by systematic screening of a blood and urine sample.

SECONDARY OUTCOMES:
The delay of detection of a cause for a first afebrile seizure in paediatric patients. | Day 1
  It is the time between the admission to paediatric emergency unit and the detection of the first afebrile seizure's cause for paediatric patients
The length of stay in Toulouse paediatric emergency unit or in hospitalization. | Day 1
number of tests performed in the search of an aetiology | Day 1
The number of tests performed in the search of an aetiology. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Claudet, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Hôpital des enfants, Toulouse, Midi-Pyrénées, France

REFERENCES:
- [Background] Bartoli M, Berny C, Danel V, Delahaye A, Desch G, Guitton J, Lacarelle B, Lapostolle F, Mathieu D, Megarbane B, Nisse P, Szymanowicz A, Capolaghi B; Toxicology and Clinical Biology Working Group. [Recommendations for the prescription, implementation and interpretation of medical examinations in biology in the context of severe poisoning]. Ann Biol Clin (Paris). 2012 Jul-Aug;70(4):431-50. doi: 10.1684/abc.2012.0726. French. PMID 22796615
- [Background] Hauser WA, Beghi E. First seizure definitions and worldwide incidence and mortality. Epilepsia. 2008;49 Suppl 1:8-12. doi: 10.1111/j.1528-1167.2008.01443.x. PMID 18184148
- [Background] Chelse AB, Kelley K, Hageman JR, Koh S. Initial evaluation and management of a first seizure in children. Pediatr Ann. 2013 Dec;42(12):244-8. doi: 10.3928/00904481-20131122-08. PMID 24295157
- [Background] Finkelstein Y, Hutson JR, Freedman SB, Wax P, Brent J; Toxicology Investigators Consortium (ToxIC) Case Registry. Drug-induced seizures in children and adolescents presenting for emergency care: current and emerging trends. Clin Toxicol (Phila). 2013 Sep-Oct;51(8):761-6. doi: 10.3109/15563650.2013.829233. Epub 2013 Aug 19. PMID 23957582
- [Background] Thundiyil JG, Kearney TE, Olson KR. Evolving epidemiology of drug-induced seizures reported to a Poison Control Center System. J Med Toxicol. 2007 Mar;3(1):15-9. doi: 10.1007/BF03161033. PMID 18072153
- [Background] Reichert C, Reichert P, Monnet-Tschudi F, Kupferschmidt H, Ceschi A, Rauber-Luthy C. Seizures after single-agent overdose with pharmaceutical drugs: analysis of cases reported to a poison center. Clin Toxicol (Phila). 2014 Jul;52(6):629-34. doi: 10.3109/15563650.2014.918627. Epub 2014 May 20. PMID 24844578
- [Background] Thundiyil JG, Rowley F, Papa L, Olson KR, Kearney TE. Risk factors for complications of drug-induced seizures. J Med Toxicol. 2011 Mar;7(1):16-23. doi: 10.1007/s13181-010-0096-4. PMID 20661684
- [Background] Citak A, Soysal DD, Ucsel R, Karabocuoglu M, Uzel N. Seizures associated with poisoning in children: tricyclic antidepressant intoxication. Pediatr Int. 2006 Dec;48(6):582-5. doi: 10.1111/j.1442-200X.2006.02276.x. PMID 17168978
- [Background] Sharma AN, Hoffman RJ. Toxin-related seizures. Emerg Med Clin North Am. 2011 Feb;29(1):125-39. doi: 10.1016/j.emc.2010.08.011. PMID 21109109
- [Background] Chen HY, Albertson TE, Olson KR. Treatment of drug-induced seizures. Br J Clin Pharmacol. 2016 Mar;81(3):412-9. doi: 10.1111/bcp.12720. Epub 2015 Sep 17. PMID 26174744
- [Background] Cerminara C, El-Malhany N, Roberto D, Lo Castro A, Curatolo P. Seizures induced by desloratadine, a second-generation antihistamine: clinical observations. Neuropediatrics. 2013 Aug;44(4):222-4. doi: 10.1055/s-0033-1333871. Epub 2013 Mar 1. PMID 23456992